CLINICAL TRIAL: NCT05813093
Title: Interleaved TMS-fMRI to Evaluate Intermittent Theta-burst and Dorsolateral Prefrontal Circuit Engagement in Ultra-treatment Resistant Depression
Brief Title: Interleaved TMS-fMRI in Ultra-treatment Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Sean Michael Nestor, Clinician Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5408
Record Dates: First submitted 2023-03-13; First posted 2023-04-14 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: We propose a pilot study using state-of-the-art concurrent fMRI acquisition to identify circuits involved with mood, and to subsequently use concurrent interleaved iTBS-fMRI and neuronavigation to examine/dynamically probe, for the first time, how iTBS of the left DLPFC mediates target engagement/functional connectivity between the DLPFC-sgACC circuit and reward system in TRD versus UTRD across varying stimulation amplitude (i.e. doses). Our secondary objective is to identify subtypes of UTRD/TRD patients from pre-treatment iTBS-fMRI who demonstrate clinical improvement in depressive symptoms with a previously validated accelerated iTBS treatment protocol over 5 consecutive days [6].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Accelerated iTBS treatment (Experimental): accelerated iTBS treatment protocol over 5 consecutive days
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Accelerated iTBS treatment

SUMMARY:
This is a study that will recruit patients from the neurosurgery clinic and the regular TMS clinic. It's a smaller study designed to collect brain imaging pre-treatment and then use image guided TMS to treat patient with a one week "accelerated" rTMS protocol using the research TMS machine that is housed in Dr. Sean Nestor's lab. The idea is to examine whether severe treatment resistant depression has a different brain signature than less severe/TRD and whether the investigators can get a therapeutic response from patients that would otherwise undergo neurosurgery or will ultimately undergo neurosurgery.

DETAILED DESCRIPTION:
The objective of this study is to assess plasticity in both whole brain connectivity and a mood/affective circuit involving the dorsolateral prefrontal cortex (DLPFC) in individuals undergoing repetitive transcranial magnetic stimulation (rTMS) for treatment of ultra-treatment resistant depression. Our second aim is to explore how these markers predict response to rTMS. The DLPFC is a brain region known to support mood regulation and has functional brain activity that is altered in depression. Past evidence from healthy controls suggests that rTMS increases coupling of the DLPFC network with another functional brain network involved in reward. Using sophisticated neuroimaging techniques that concurrently capture functional MRI while patients are being stimulated with rTMS, the investigators will identify patterns of brain activity associated with depressed mood and measure the coupling of the DLPFC mood circuit with a reward network prior to an acute course of rTMS. Following baseline imaging, all patients will then undergo an accelerated rTMS protocol over the course of five days, using the pre-treatment imaging to localize the brain region (circuit) targeted by the TMS coil. The investigators will also use questionnaires to assess mood and function before, during and after rTMS treatment. Two comparison groups will be included in this study: 1) patients with depression who have ultra-treatment resistant depression and have been referred for consideration of neurosurgical neuromodulation for depression, and 2) persons with milder treatment resistant depression who are referred to the Harquail Centre for rTMS treatment of depression. This research will help us better understand the mechanisms of how rTMS modulates brain activity, improve TMS targeting in depression, and identify pre-treatment imaging that predict response to rTMS with potentially far-reaching clinical implications.

ELIGIBILITY:
Inclusion criteria:

* Age 20-65
* Have a diagnosis of MDD or persistent depressive disorder and meet criteria for a major depressive episode (moderate-severe) according to the DSM 5.0 with a 17-item Hamilton Rating Scale Score in Depression (HRSD-17) of >=18
* UTRD subjects will also have a duration of depressive symptoms >=5 years, treatment resistance to antidepressants will be defined by Maudsley-staging, failing >6 antidepressants (level 4) and >1 adjunctive antidepressants of adequate dose/duration, failed at >=1 psychotherapy, and no response to >=1 trial of esketamine, IV ketamine, ECT or rTMS
* Milder TRD participants will have failed at least 1 antidepressant medication of adequate dose/duration and never had neuromodulation treatment

Exclusion criteria:

* Contraindications to MRI
* Medical/psychiatric co-morbidities that prevent participation in the study or where depression is not the primary psychiatric symptom of concern
* History of psychosis, pregnancy, substance dependence within the last 6 months
* Active neurological disorder
* History of seizure disorder
* Cognitive impairment
* Unable to provide informed consent on their own
* Pregnant

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-07-07 (Estimated); Study Completion 2025-07-07 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptomatology | 3 years
  Change in depression symptomatology as assessed by the clinician-rated 17-item Hamilton Depression Rating Scale (range 0-52)
Imaging | 3 years
  fMRI target engagement in the subgenual anterior cingulate cortex (sgACC)

OTHER OUTCOMES:
Predictive capacity of fMRI target engagement | 3 years
  Prognostic value of target engagement in the sgACC (active - sham) in predicting response and remission, above and beyond readily-available clinical and demographic variables (age, sex, baseline depression severity, number of prior treatments in current depressive episode). This will be assessed via AUC of the model(s) in predicting outcomes and by comparing the fit of models with and without sgACC target engagement (t-statistic from ROI analysis based on Freesurfer anatomical mask for bilateral sgACC) to test for significant improvement orthogonal to readily-available clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No